CLINICAL TRIAL: NCT00968370
Title: Randomized, Controlled Clinical Trial of Day-care Based and Hospitalized Management of Severe and Very Severe Pneumonia, With Severe Malnutrition, With/Without Associated Co-morbidities in Children
Brief Title: Trial in Childhood Pneumonia With Malnutrition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Basel (Other); Institute of Child health & Shishu Sasthya Foundation Hospital (ICHSH), Bangladesh (Unknown); Radda MCH-FP Centre, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-009
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2009-08

CONDITIONS: Malnutrition; Pneumonia
Keywords: Severe and very severe pneumonia; severe malnutrition; children; day-care management; hospital management
MeSH Terms: conditions — Malnutrition; Pneumonia | interventions — Hospital Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Day-care clinic (Active Comparator): Inj. Ceftriaxone and other micronutrients will be given to children at the day-care clinic from 8:00 a.m. to 5:00 p.m. daily.
  Interventions: Other: Day-care clinic
- Hospital management (Other): Hospital management: all children admitted at the hospital will be managed with injection Ceftriaxone and other micronutrients for the total duration of hospitalization as per approved protocol.
  Interventions: Other: Hospital Management

INTERVENTIONS:
Other: Day-care clinic — Inj. Ceftriaxone and other micronutrients will be given to children at the day-care clinic from 8:00 a.m. to 5:00 p.m. daily.
  Arms: Day-care clinic
Other: Hospital Management — Inj. Ceftriaxone and other micronutrients will be given to children at the hospital from admission till discharge.
  Arms: Hospital management

SUMMARY:
The impetus for this study came from the findings of the investigators' recently published study entitled "Day-care management of severe and very severe pneumonia, without associated co-morbidities such as severe malnutrition, in an urban health clinic in Dhaka, Bangladesh". If day-care management is found to have comparable efficacy to that of hospital management of severe and very severe pneumonia in children then they could be managed at outpatient, day-care set ups reducing hospitalization and thus freeing beds for management of other children who need hospital care. Such management could also be implemented in rural areas of Bangladesh and potentially to other developing countries. Additionally, availability of the treatment facility in community set-ups will be cost and time saving for the population. But, as patients with severe malnutrition were excluded from the pilot study for ethical reasons, the peer reviewers of the manuscript felt that the study findings cannot be applied to the treatment of severe and very severe pneumonia in general. Similarly, management of severely malnourished children with associated complications relies on hospital-based treatment. In another study, a day-care clinic approach by providing antibiotics, micronutrients, diet and supportive care to severely malnourished children showed that they could be successfully managed at existing day-care clinics using a protocolized approach. Therefore, after the successful conduction and publication of these two study results in international journals with severe and very severe pneumonia as well as severe malnutrition at the day-care clinic, it is mandatory to perform the final study where the investigators will include severe malnutrition as well as associated co-morbidities to be applied to the treatment of severe and severe pneumonia in children in general to make the treatment approach more widely applicable.

DETAILED DESCRIPTION:
Acute lower respiratory infections particulary pneumonia, are the leading cause of childhood morbidity and death in the developing countries such as Bangladesh [3]. Acute respiratory tract infection causes more than 2 million child deaths worldwide each year, mostly from pneumonia and 90% of them occur in less-developed countries [4-6]. Recent estimates suggest that 1.9 million (95% CI 1.6 million to 2.2 million) children died from acute respiratory tract infection throughout the world in 2000, and 70% of them occurred in Africa and Southeast Asia [7]. ARI is also a major cause of visits to the outpatient and emergency departments as well as admissions to the hospitals. Although bronchiolitis, tracheobronchitis and pneumonia, each accounts for about one-third of ALRI cases, pneumonia is responsible for most ALRI deaths. Three studies that reported diagnoses in children who died of ALRI revealed that a median of 89% (range 71% to 100%) of ALRI deaths was associated with pneumonia [8-10]. In Bangladesh, acute lower respiratory tract infections account for 25% of deaths in the under-5 age group and 40% of all infantile deaths [11]. A study conducted at the Dhaka Hospital of ICDDR,B in 1986-88 in 401 under-5 children with ALRI has documented that pneumonia was most common among them and a respiratory pathogen (both bacterial and viral) was identified in 30% cases. The case fatality rates were 14% in bacterial pneumonia and 3% in viral pneumonia [12]. Bacterial infections play a major role in childhood pneumonia in developing countries. Pooled data from lung aspiration studies, mostly from developing countries, reported bacterial isolation rates of 52-62% [13, 14]. The case-fatality rate in severe ALRI in children aged 1-4 years was reported to be 10-15 times higher in the developing than in the developed countries [15, 16]. It is usually not possible to determine the specific cause of pneumonia by either clinical or chest X-ray features. In children, Streptococcus pneumoniae and Haemophilus influenzae are the two most important bacterial pathogens [17, 18]. Respiratory Syncytial Virus (RSV) is also an important cause of ARI among preschool children [12, 18]. Emerging evidence suggests that Mycoplasma pneumoniae and Chlamydia pneumoniae may cause pneumonia among older children. Available data also suggests that mixed viral and bacterial infections are common in children in developing countries [12], which require antimicrobial therapy. The WHO recommendations for treatment of pneumonia are based on data that Streptococcus pneumoniae and Haemophilus influenzae are the most common causes of bacterial pneumonia in developing countries [9].

Depending on clinical presentation, pneumonia can be classified as very severe, severe or non-severe, with specific treatment guidelines available for each [8, 16, 19, 20]. The WHO defines very severe pneumonia as clinical symptoms and signs of pneumonia (cough or difficulty breathing with one or more danger signs like cyanosis, convulsions, drowsiness, stridor in calm child or inability to drink, all signifying hypoxaemia or severe respiratory distress) and severe clinical malnutrition [8, 16, 19, 20]. Severe pneumonia is defined as cough or difficulty breathing with lower chest wall in drawing with or without fast breathing defined as the respiratory rate ³ 50 breaths per minute for children aged 2-11 months and ³ 40 breaths per minute for children aged 12-59 months [8, 16, 19, 20]. Lower chest wall in drawing is defined as inward movement of the bony structures of the lower chest wall with inspiration, observed while the child is at rest [21]. Finally, non-severe pneumonia is defined as cough or difficulty breathing with fast breathing as defined earlier [8, 16, 19, 20]. Antibiotic therapy is indicated irrespective of the severity of pneumonia. Proper management of children presenting in health centres and hospitals with respiratory symptoms is the cornerstone of acute respiratory infection control. To address the high mortality associated with ALRI, WHO launched a programme for control of ARI with the major objective to reduce the child mortality and to promote rational use of antibiotic. Current standard ARI case management recommends ambulatory treatment of children with cough and normal breathing without antibiotics assuming viral infection or mild bacterial infections; treatment of those with rapid respiration (tachypnoea) indicating lower respiratory infection or pneumonia with an antibiotic (non-severe pneumonia); and hospitalisation of those with lower chest wall in drawing (indicative of severe pneumonia) and treatment with parenteral antibiotics and supportive cares [22, 23]. Vaccination against measles, pertussis, Haemophilus influenzae type b (Hib) and Streptococcus pneumoniae can help decrease the incidence and/or lessen the severity of respiratory infections. However, newer vaccines against respiratory infections such as Hib and pneumococcal conjugate vaccines are not widely available in developing countries. Under-5 children with respiratory symptoms are brought to the general practitioners as well as to primary health care facilities for treatment and health care providers are required to differentiate between acute upper respiratory infections (AURI) and acute lower respiratory infections (ALRI)/pneumonia, categorize severity of pneumonia taking into consideration the nutritional status of the patients, and provide either ambulatory therapy or refer patients for hospitalization, as appropriate.

Management of severe and very severe pneumonia in children relies on hospital-based treatment, but practical barriers often prevent children in areas with highest rates from receiving hospital care. It is recommended that children with severe or very severe pneumonia be hospitalised [8, 16, 19, 20] for supportive treatment, including suction, oxygen therapy for hypoxemia, fluid and nutritional management, and close monitoring [8, 16, 19, 20]. In Bangladesh, there are not enough hospital beds for admission of all severe and very severe cases of pneumonia. In addition, hospitalization may not be possible because of the inability of parents to visit the hospital. Reliable demographic information on this issue is not available in most hospitals in Bangladesh due to poor record keeping system. However, we have reviewed data for a 2-month period (May and June 2007) from the Institute of Child Health and Shishu Sasthya Foundation Hospital (ICHSH), Mirpur, Dhaka, and observed that only 52/120 (43%) children with severe and very severe pneumonia were admitted into the hospital, and the majority (57%) could not be admitted due to the lack of beds and most of them were sent home after some supportive therapy and parenteral antibiotics from the outpatient department of the hospital. It is therefore important to provide institutional care for children who cannot be hospitalised. A prospective observational study was conducted to examine the feasibility of day-care-facility-based, modified primary care as an alternative for children denied hospital admission who would otherwise be sent home. We developed and prospectively evaluated a day-care clinic approach of management by providing antibiotics, feeding and supportive care during stay at the clinic, and continuation of care at home by parents as an effective alternative to hospitalization for such children. We have recently published the study results as "Day-care management of severe and very severe pneumonia, without associated co-morbidities such as severe malnutrition, in an urban health clinic in Dhaka, Bangladesh [1]". From June 2003 to May 2005, 251 children with severe and very severe pneumonia were enrolled at the Radda Clinic. The mean±SD age of the children was 7 ±7 months, and 143/251 (57%) of them were hypoxemic with mean ± SD oxygen saturation of 93 ± 4% that increased to 98 ± 3% on oxygen therapy. The mean ± SD day-care period was 7 ± 2 days. Day-care management of severe and very severe pneumonia was assessed successful in 234/251 [93% (95% CI, 89-96%)] children, and the management was assessed to have failed in the remaining 17/251 [7% (95% CI, 4.3-10.6%)] children of whom 11/251 [4.4% (95% CI, 2.5-7.7%)] had to be referred to hospital and 6/251 [2.4% (95% CI 1.1-5.1%)] discontinued treatment. There were no deaths during the day-care study period; however, 4/251 [1.6% (95% CI 0.6%-4%)] children died during the 3-month follow-up period, and another 11/251 [4.4% (95% CI, 2.5-7.7%)] required hospital admission during the 3-months' follow-up period. The results of the study indicate that children with severe and very severe pneumonia without associated co-morbidities such as severe malnutrition can be successfully managed at day-care clinics [1]. If the day-care management is found to have comparable efficacy to that of hospitalized management of severe and very severe pneumonia in children then they could be managed at day-care set ups on an outpatient basis, reducing hospitalization and thus freeing up of beds for management of other children with greater need for hospital care. Additionally, availability of the treatment facility in community set-ups will be both time-and cost-savings for the population. But, as patients with severe malnutrition were excluded from the pilot study for ethical reasons, the peer journal reviewers [1] correctly commented that the study findings cannot be generalised and applied to the treatment of severe and very severe pneumonia.

Similarly, the case-fatality from severe malnutrition has been as high as 60% in the 1990's primarily due to faulty case management [24-26]. The management of severely malnourished children with associated complications relies on hospital-based treatment. In Bangladesh, only a few hospitals have beds dedicated for the management of severely malnourished children. Hospitalization may not also be possible as a result of the inability of the parents to visit a hospital either due to distance or financial reason (s), even after appropriate referral. It is, however, important to provide institutional care to such children, at least until stabilization of their acute conditions. If such children are sent home with antibiotics, it would be important to establish an expensive, home follow up system, without which a significant proportion of them could be reasonably expected to have a fatal outcome. With the implementation of a protocolised management at the Dhaka Hospital, ICDDR,B, the case-fatality of such children reduced from 19% to 5% [27, 28]. In another study, we evaluated a day-care clinic approach of management of severely malnourished children by providing antibiotics, micronutrients, diet, and supportive care during stay at an established day-care centers, followed by continuation of care by parents at home as an effective alternative to hospitalization. From February 2001 to November 2003, 264 severely malnourished children were enrolled at the Radda Clinic, where they received protocolized management with antibiotics, micronutrients and milk-based diet from 08:00 to 17:00 daily, while their mothers were educated on continuation of supportive care at home at night. They were transitioned to the day-care nutrition rehabilitation unit (NRU) of the Radda Clinic following resolution of acute illness, received NRU diets daily until attainment of 80% weight-for-length. Fifty-two percent of the children were boys, and 78%, 21% and 1% of all children had marasmus, marasmus-kwashiorkor and kwashiorkor, respectively. Only 13% had severe malnutrition alone, while 35% had pneumonia, 35% had diarrhoea and 17% had both pneumonia and diarrhoea. The mean ± SD duration of acute and NRU phases were 8 ± 4 and 14 ± 13 days respectively. The mean ± SD weight gain (g/kg) of the children was more rapid during acute (10 ± 7) than the NRU phase (6 ± 5). The day-care management of severe malnutrition was assessed successful in 216/264 [82% (95% CI, 77-86%)] children, and failure in the remaining 48/264 [18% (95% CI, 14-23%)] children of whom 17/264 [6% (95% CI, 4-10%)] had to be referred to hospital and 31/264 [12% (95% CI, 8-16%)] discontinued treatment. The results clearly demonstrated that severely malnourished children could be successfully managed at existing day-care clinics using a protocolized approach [2].

Therefore, after the successful conduction and publication of results of these two studies on management of severe and very severe pneumonia [1] and severe malnutrition [2] at the day-care clinic, it is prudent to perform the final study in which we will assess if treatment of children with severe and very severe pneumonia in association with severe malnutrition will be possible on a day-care basis. If successful, this treatment approach could be more widely applicable. In the proposed study, we would identify under-5 children with severe and very severe pneumonia with severe malnutrition with/without associated co-morbidities attending the outpatient department of the Radda Clinic and the outpatient and emergency departments of ICHSH and randomize them, in equal numbers, for management either at the day-care centre (Radda Clinic) or hospital (ICHSH), subject to the consent of respective parents/guardians. About 3000 children with pneumonia visit the Radda Clinic each year, and we estimate that about 200 of them will have severe and very severe pneumonia with severe malnutrition requiring hospitalization. Similarly, about 700 children with severe and very severe pneumonia with severe malnutrition visit the outpatient and emergency departments of the ICHSH each year. Our study patients will be selected from these children population of the Radda Clinic and ICHSH, and we hope to complete enrolment of the requisite 440 (220/site) children during 3-year period of the study.

Rationale

Malnutrition and severe malnutrition are prevalent and ALRI/pneumonia is the leading cause of under-5 morbidity and deaths in Bangladesh. Hospital management is recommended for children with either or both of these problems. However, there simply is not enough beds to hospitalise every child with these problems. It is often not possible to provide appropriate treatment and supportive care at home to children refused admission to a hospital. With a few exceptions, childhood malnutrition is a problem of the poor, and thus parents of children with severe malnutrition and/or pneumonia are often unable to provide private care to their children, and some times unable to take their children to a hospital far off from their community. What happens to such children remains largely unknown; however, many can be expected to have a fatal outcome. Successful management of such children at a day-care clinic in their community would provide better access to their treatment and care and affordable to the parents. Proved effective, this management could also be implemented in Bangladesh and potentially to other developing countries. The day-care based management is expected to be cost effective intervention and contribute significantly to reduction of under-5 child mortality due to severe and very severe pneumonia as well as severe malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 to 59 months
* Sex: Both boys and girls
* Severe and very severe pneumonia
* Severe malnutrition (defined as < - 3 weight-for-height Z-score)
* Attending Radda Clinic or ICHSH between 8:00 to 16:00
* Written informed consent by respective parents/guardians

Exclusion Criteria:

* Non-severe pneumonia
* Nosocomial pneumonia
* Bronchiolitis
* Bronchial asthma
* Living long distance (>5 km) from the Radda Clinic and ICHSH
* Visits during late hours of the day (after 16:00)
* Parents/guardians not consenting for enrolment of children in the study

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Actual)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proportion of success with 95% confidence interval (CI) | 3 years

SECONDARY OUTCOMES:
Case fatality rate with 95% CI -day-care clinic/hospital | 3 years
Proportion of failure rate with 95% CI | 3 years
Duration of illness (d) | 3 years
Proportion of referral & discontinuation with 95% CI | 3 years
Duration of success (d) | 3 years
Development of complications | 3 years
Cost of treatment | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Ashraf H, Alam NH, Sultana M, Jahan SA, Begum N, Farzana S, Chisti MJ, Kamal M, Shamsuzzaman A, Ahmed T, Khan JAM, Fuchs GJ, Duke T, Gyr N. Day clinic vs. hospital care of pneumonia and severe malnutrition in children under five: a randomised trial. Trop Med Int Health. 2019 Jul;24(7):922-931. doi: 10.1111/tmi.13242. Epub 2019 May 14. PMID 31046165